CLINICAL TRIAL: NCT07147140
Title: Evaluation of Physiological Parameters in Patients With Complex Regional Pain Syndrome of the Lower Limbs Treated With Dorsal Root Ganglion Stimulation.
Brief Title: Physiological Parameters in CRPS Patients Treated With Dorsal Root Ganglion Stimulation
Acronym: EPIC-DRG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AZ Delta (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANE 20241129
Record Dates: First submitted 2025-04-14; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-04

CONDITIONS: CRPS (Complex Regional Pain Syndrome) Type I
Keywords: Complex regional pain syndrome type 1; dorsal root ganglion stimulation; automonic outcome parameters
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of cessation dorsal root ganglion stimulation in patients with CRPS I. (Experimental)
  Interventions: Device: dorsal root ganglion stimulation cessation

INTERVENTIONS:
Device: dorsal root ganglion stimulation cessation — Treatment of DRGS will be stopped at home and physiological parameters will be monitored with bio wearables at home. physiological parameters will be monitored during a baseline period, before stopping DRGS. While DRGS is stopped. And during the period while the DRGS is turned back on.

SUMMARY:
1. Objective and Rationale: The study seeks to evaluate how Dorsal Root Ganglion Stimulation (DRGS) influences autonomic functions in patients suffering from Complex Regional Pain Syndrome type I (CRPS I), offering new metrics beyond pain scores to assess therapeutic efficacy.
2. Innovative Approach: Continuous monitoring of patients using validated, CE-marked biosensors (Corsano Biosensor and Motionwatch8) to collect real-time physiological data during active DRGS therapy and therapy cessation periods.
3. Clinical Impact: Results from this study may improve patient management strategies and refine treatment protocols for individuals living with CRPS I.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Complex Regional Pain Syndrome Type I (CRPS I) of the lower limbs.
* Currently treated with Dorsal Root Ganglion Stimulation (DRGS).
* Patients must experience > 50% pain relief with DRGS therapy for at least three months.
* Willingness and ability to comply with the study requirements, including wearing biosensors, and sharing their physiological parameters.

Exclusion Criteria:

* Refusal or inability to wear biosensor wearables.
* Current pregnancy.
* Patients with other significant medical conditions that could affect autonomic function.
* Known allergies or intolerance to materials used in biosensors.
* Diagnosis of untreated Obstructive Sleep Apnea Syndrome (OSAS).
* Ongoing psychiatric disorders

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | 1 week
  Heart Rate (beats per minute), measured using the Corsano Biosensor 287-2 wearable device (CE-MDR certified)
Heart Rate Variability | 1 week
  Heart Rate Variability (milliseconds), measured using the Corsano Biosensor 287-2 wearable device (CE-MDR certified)
Respiratory Rate | 1 week
  Respiratory Rate (breaths per minute), measured using the Corsano Biosensor 287-2 wearable device (CE-MDR certified)
Blood Pressure | 1 week
  Non-invasive Cuffless Blood Pressure: systolic, mean and diastolic (mmHg), measured using the Corsano Biosensor 287-2 wearable device (CE-MDR certified)
Body Temperature | 1 week
  Core Body Temperature (°C), measured using the Corsano Biosensor 287-2 wearable device (CE-MDR certified)
Oxygen Saturation | 1 week
  Oxygen Saturation (SpO2, %), measured using the Corsano Biosensor 287-2 wearable device (CE-MDR certified)
Sleep Quality | 1 week
  Sleep quality is measured using the MotionWatch 8 actigraphy device (FDA-cleared, CE-marked). For each night of sleep, the bed times and get-up times are entered (either manually, graphically or automatically) and the software automatically determines the sleep start and end times. The analysis then utilises the night-time movement data (e.g. immobile mins and mobile mins) to determine the quality of sleep and provides a list of key sleep parameters.
Physical Activity | 1 week
  Physical Activity (activity counts per time frame) is measured using the MotionWatch 8 actigraphy device (FDA-cleared, CE-marked).

SECONDARY OUTCOMES:
Pain intensity | 1 week
  Pain intensity (patient-reported) will be assessed using the Numeric Rating Scale (NRS; 0 = no pain, 10 = worst possible pain), recorded three times daily.
Sleep quality | 1 week
  Sleep quality (patient-reported) will be evaluated with a five-point Likert scale (1 = strongly disagree to 5 = strongly agree) based on specific sleep-related statements.
Patient Global Impression of Improvement | 1 week
  Patient Global Impression of Improvement (PGI-I) will be used to assess overall patient-perceived change, using a seven-point Likert scale (1 = very much improved, 7 = very much worse).
Pain condition-related medication usage | 1 week
  Medication intake will be recorded daily by the participant as a count of analgesic medication dosages taken.

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Delta, Roeselare, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Plan Description:
  De-identified individual participant data (IPD), including physiological parameters (heart rate variability, respiratory rate, blood pressure, oxygen saturation, skin temperature) and secondary outcomes (pain intensity scores, sleep quality assessments, medication intake, and patient global impression of improvement) will be shared with the Research Stimulus Group at Vrije Universiteit Brussel. The data will be used for real-time monitoring, statistical analysis, and preparation of scientific manuscripts related to this study.
  Access Criteria:
  Access to the IPD will be restricted to members of the Research Stimulus Group who are directly involved in the analysis and interpretation of the EPIC-DRG study data. Data handling will fully comply with GDPR regulations and institutional data protection policies. No public sharing of raw data is planned.
  Time Frame:
  Data will be transmitted continuously throughout the study period to enable interim analysis and monitoring, w
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Anticipated start date 29th April 2025 and anticipated end date 31st of October 2025.
Access Criteria: Vrije Universiteit Brussel (Research Stimulus Group). They will access the data through an API provided by AZ Delta Research Center.

REFERENCES:
- [Background] Patterson DG, Wilson D, Fishman MA, Moore G, Skaribas I, Heros R, Dehghan S, Ross E, Kyani A. Objective wearable measures correlate with self-reported chronic pain levels in people with spinal cord stimulation systems. NPJ Digit Med. 2023 Aug 15;6(1):146. doi: 10.1038/s41746-023-00892-x. PMID 37582839